CLINICAL TRIAL: NCT02217241
Title: Effect of Hand-off Skills Training for Students During the Medicine Clerkship: A Randomized Study
Brief Title: Effect of Hand-off Skills Training for Students During the Medicine Clerkship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Juan Reyes, Assistant Professor of Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 101125
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Patient Handoff

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Students in the intervention group participated in a one-hour interactive, small-group handoff workshop facilitated by a study investigator. The workshop focused on the importance of specific handoff skills to patient safety.
  Interventions: Other: Handoff Workshop
- Control (No Intervention)

INTERVENTIONS:
Other: Handoff Workshop
  Arms: Intervention

SUMMARY:
The purpose of this study is to assess the effectiveness of an educational intervention on handoffs implemented during the third year of medical school. It also assesses whether these skills are maintained over time into their fourth year of training and whether there is transfer from the simulated setting into the clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* Third Year Medicine Clerks

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluate workshop effectiveness of students undergoing the intervention, rated before and after the workshop utilizing standardized cases and a validated Handoff Rating Scale. | up to 45 minutes post-intervention

OTHER OUTCOMES:
Assess durability of the training by rating intervention and control group students on a third standardized case during their fourth year AI on internal medicine. | up to 12 months after intervention
Assess the transfer of handoff skills into the clinical setting by observing AI students in both the intervention and control groups providing real-time handoffs. | Up to 12 months after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University School of Medicine; The George Washington University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Vidyarthi AR, Arora V, Schnipper JL, Wall SD, Wachter RM. Managing discontinuity in academic medical centers: strategies for a safe and effective resident sign-out. J Hosp Med. 2006 Jul;1(4):257-66. doi: 10.1002/jhm.103. PMID 17219508
- [Background] Laine C, Goldman L, Soukup JR, Hayes JG. The impact of a regulation restricting medical house staff working hours on the quality of patient care. JAMA. 1993 Jan 20;269(3):374-8. PMID 8418344
- [Background] Lofgren RP, Gottlieb D, Williams RA, Rich EC. Post-call transfer of resident responsibility: its effect on patient care. J Gen Intern Med. 1990 Nov-Dec;5(6):501-5. doi: 10.1007/BF02600880. PMID 2266432
- [Background] Horwitz LI, Krumholz HM, Green ML, Huot SJ. Transfers of patient care between house staff on internal medicine wards: a national survey. Arch Intern Med. 2006 Jun 12;166(11):1173-7. doi: 10.1001/archinte.166.11.1173. PMID 16772243
- [Background] Arora VM, Eastment MC, Bethea ED, Farnan JM, Friedman ES. Participation and experience of third-year medical students in handoffs: time to sign out? J Gen Intern Med. 2013 Aug;28(8):994-8. doi: 10.1007/s11606-012-2297-9. PMID 23595921
- [Background] Gordon M, Findley R. Educational interventions to improve handover in health care: a systematic review. Med Educ. 2011 Nov;45(11):1081-9. doi: 10.1111/j.1365-2923.2011.04049.x. Epub 2011 Sep 20. PMID 21933243
- [Background] Farnan JM, Paro JA, Rodriguez RM, Reddy ST, Horwitz LI, Johnson JK, Arora VM. Hand-off education and evaluation: piloting the observed simulated hand-off experience (OSHE). J Gen Intern Med. 2010 Feb;25(2):129-34. doi: 10.1007/s11606-009-1170-y. PMID 19924489
- [Background] Horwitz LI, Moin T, Green ML. Development and implementation of an oral sign-out skills curriculum. J Gen Intern Med. 2007 Oct;22(10):1470-4. doi: 10.1007/s11606-007-0331-0. Epub 2007 Aug 3. PMID 17674110
- [Background] Chu ES, Reid M, Schulz T, Burden M, Mancini D, Ambardekar AV, Keniston A, Albert RK. A structured handoff program for interns. Acad Med. 2009 Mar;84(3):347-52. doi: 10.1097/ACM.0b013e3181970829. PMID 19240442
- [Background] Gakhar B, Spencer AL. Using direct observation, formal evaluation, and an interactive curriculum to improve the sign-out practices of internal medicine interns. Acad Med. 2010 Jul;85(7):1182-8. doi: 10.1097/ACM.0b013e3181da8370. PMID 20375830
- [Background] Klamen DL, Reynolds KL, Yale B, Aiello M. Students learning handovers in a simulated in-patient unit. Med Educ. 2009 Nov;43(11):1097-8. doi: 10.1111/j.1365-2923.2009.03488.x. Epub 2009 Oct 3. No abstract available. PMID 19799733
- [Background] Darbyshire D, Gordon M, Baker P. Teaching handover of care to medical students. Clin Teach. 2013 Feb;10(1):32-7. doi: 10.1111/j.1743-498X.2012.00610.x. PMID 23294741
- [Background] Chu ES, Reid M, Burden M, Mancini D, Schulz T, Keniston A, Sarcone E, Albert RK. Effectiveness of a course designed to teach handoffs to medical students. J Hosp Med. 2010 Jul-Aug;5(6):344-8. doi: 10.1002/jhm.633. PMID 20803673
- [Background] Starmer AJ, Sectish TC, Simon DW, Keohane C, McSweeney ME, Chung EY, Yoon CS, Lipsitz SR, Wassner AJ, Harper MB, Landrigan CP. Rates of medical errors and preventable adverse events among hospitalized children following implementation of a resident handoff bundle. JAMA. 2013 Dec 4;310(21):2262-70. doi: 10.1001/jama.2013.281961. PMID 24302089
- [Background] Curtis JR, Back AL, Ford DW, Downey L, Shannon SE, Doorenbos AZ, Kross EK, Reinke LF, Feemster LC, Edlund B, Arnold RW, O'Connor K, Engelberg RA. Effect of communication skills training for residents and nurse practitioners on quality of communication with patients with serious illness: a randomized trial. JAMA. 2013 Dec 4;310(21):2271-81. doi: 10.1001/jama.2013.282081. PMID 24302090
- [Derived] Reyes JA, Greenberg L, Amdur R, Gehring J, Lesky LG. Effect of handoff skills training for students during the medicine clerkship: a quasi-randomized study. Adv Health Sci Educ Theory Pract. 2016 Mar;21(1):163-73. doi: 10.1007/s10459-015-9621-1. Epub 2015 Jul 15. PMID 26174046